CLINICAL TRIAL: NCT05079425
Title: A Randomized, Double-blind, Placebo-controlled, Single and Multiple Ascending Dose Phase 1 Clinical Trial to Evaluate Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Food Effect After the Oral Administration of NXC736 in Healthy Male Subjects
Brief Title: A First-in-Human Study to Assess Single and Multiple Doses of NXC736 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NEXTGEN Bioscience (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Other
Other Study IDs: NXC736-001
Record Dates: First submitted 2021-09-27; First posted 2021-10-15 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part A: Fasting (Experimental): Single ascending dose (SAD).
  Interventions: Drug: NXC736; Drug: Placebo
- Part A: Fed (Experimental): Single ascending dose (SAD).
  Interventions: Drug: NXC736; Drug: Placebo
- Part B: Fasting (Experimental): Multiple Ascending Dose (MAD)
  Interventions: Drug: NXC736; Drug: Placebo

INTERVENTIONS:
Drug: NXC736 — Oral administration
Drug: Placebo — Oral administration

SUMMARY:
This is a randomized, double-blind, placebo- controlled, single and multiple dosing, dose-escalation clinical phase 1 trial to investigate the safety, tolerability, pharmacokinetics and pharmacodynamics of NXC736 after oral administration in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males aged between 19 and 55 at screening
* Those whose weight is between 55 and 90 kg and BMI is between 18.0 and 30.0
* Those who are adequate to be subjects in this study upon judgment of the investigator after physical examination, clinical laboratory test, examination by interview, etc
* Signed informed consent form

Exclusion Criteria:

* Those who have clinical significant liver, kidney, nervous system, respiratory, endocrine, hematology and oncology, cardiovascular, urinary, and mental diseases or past history
* Those who have gastrointestinal diseases or past history of gastrointestinal diseases that may affect safety and pharmacokinetic/pharmacodynamic evaluation of study drug, and those who have past history of gastrointestinal surgery (however, except simple appendectomy and herniotomy)
* A person who shows any of the following results in vital signs at the time of screening

  * Systolic blood pressure below 90 mmHg or above 140 mmHg
  * diastolic blood pressure less than 50 mmHg or greater than 90 mmHg
  * Pulse rate less than 50 beats per minute or more than 90 beats per minute
* A person who exhibits any of the following results from a 12-lead ECG test at the time of screening:

  * PR > 210 msec
  * QRS complex > 120 msec
  * QTcB > 450 msec
* A person who exhibits any of the following results in a clinical laboratory examination at the time of screening ;

  * glomerular filtration rate (eGFR, CKD-EPI) < 60 mL/min/1.73 m2
  * WBC count < 3500/μL
  * Absolute neutrophil count (ANC) < 1500/μL
  * AST/ALT > 1.5 X ULN
* Those who have a history of tuberculosis infection or who have confirmed positive tuberculosis infection as a result of the Quantiferon TB-Gold test and Chest X-ray performed at the screening test
* Persons with acute infectious diseases including herpes virus infection, herpes simplex, and herpes zoster

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | Day 49
Number of Participants with Serious Adverse Events (SAEs) | Day 49
Number of Participants with Vital Sign Abnormalities | Day 49
Number of Participants with Electrocardiogram (ECG) Abnormalities | Day 49
Number of Participants with Clinical Laboratory Abnormalities | Day 49

CONTACTS AND LOCATIONS:
Overall Officials: Seungwhan Lee, Principal Investigator — Seoul National University College of Medicine and Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No